CLINICAL TRIAL: NCT06398574
Title: Effect of Dry Needling Technique on Shoulder Muscle Functionality in Subjects With and Without Shoulder Pain.
Brief Title: Effects of Dry Needling on the Behavior of the Shoulder Muscles
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Prof. Dr. Daniel Pecos Martín, Professor, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEID/2024/1/004
Record Dates: First submitted 2024-05-01; First posted 2024-05-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Shoulder Pain
Keywords: Dry needling; Shoulder muscle strength; Surface electromyography
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real dry needling (Experimental): With the subject lying supine, a dry needling technique will be applied to the infraspinatus muscle.
  Interventions: Other: Real dry needling
- Sham dry needling (Sham Comparator): With the subject lying supine, a sham dry needling technique will be applied to the infraspinatus muscle, simulating the real procedure.
  Interventions: Other: Sham dry needling

INTERVENTIONS:
Other: Real dry needling — With the subject lying supine, a dry needling technique will be applied to the infraspinatus muscle. First, the most hyperalgesic point in the muscle will be located. Subsequently, Hong's fast-in and fast-out technique will be applied. Ten incisions will be made
  Arms: Real dry needling
Other: Sham dry needling — With the subject lying supine, a sham dry needling technique will be applied to the infraspinatus muscle. First, the most hyperalgesic point in the muscle will be located. Subsequently, Hong's fast-in and fast-out technique will be applied. Ten incisions will be made, simulating the real technique
  Arms: Sham dry needling

SUMMARY:
The main objective of this study will be to evaluate the effects of the application of the dry needling technique on the activity of the rotator cuff muscles in the shoulder.

The evaluation of the effects of the application of the dry needling technique will be carried out in subjects with and without shoulder pain.To do this, muscle strength, possible thickness changes in the muscle and electromyographic activity will be measured before and immediately after the application of a dry needling technique.

Likewise, other variables will be measured such as the pressure pain threshold (PPT), pain with a Numeric Verbal Scale, kinesiophobia and catastrophism, the shoulder pain and disability index (SPADI) and the influence of expectations about dry needling.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of legal age
* Subjects without shoulder pain or with unilateral shoulder pain of > 3 months duration.
* Have shoulder mobility of 90º of abduction and at least 30º of glenohumeral external rotation.

Exclusion Criteria:

* Have neck pain.
* Whiplash
* Having had trauma to the shoulder.
* Having fibromyalgia.
* Be pregnant.
* Being afraid of needles.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-03-20 (Estimated)

PRIMARY OUTCOMES:
Muscle strength | Change from Baseline at 15 minutes.
  The isometric strength will be assessed using a handheld dynamometer (Hand held dynamometer, MicroFET3; Hoggan Health Industries Inc.). The strength measures will included external rotation at 90° abduction in the prone position. The dynamometer will be placed just proximal to the just proximal to the styloid process of the wrist joint. Subjects will be asked to produce a 5-second maximal contraction. Muscular strength will be measured in kilograms

SECONDARY OUTCOMES:
Muscle function | Change from Baseline at 15 minutes.
  Muscle function will be measured by an ultrasound scanner with a linear transducer with a frequency range of 6-16MHz (X6-16L, 5cm footprint) will be used. The unit of measurement used will be millimeters. Muscle thickness at rest and contraction will be measured. On the other hand, the percentage of change in thickness will be measured using the equation (Contraction thickness - Rest thickness) * 100 / Rest thickness.
Shoulder Pain | Change from Baseline at 15 minutes.
  Pain intensity will be measured using the Visual Analog Scale (VAS) for pain. The VAS is a 100-mm line, oriented horizontally, with one end representing "no pain" and ten the other end representing "worst pain." Subjects will be asked to rate their current pain with a mark on the scale.
Disability | Change from Baseline at 15 minutes.
  Disability will be measured by Shoulder Pain and Disability Index (SPADI).The Spanish version of SPADI has high test-retest reliability (ICC 0.89-0.93).The clinically important minimum difference varies between 8 and 13.2. The minimum value is 0 and de maximum value is 100
Pressure Pain Threshold (PPT) | Change from Baseline at 15 minutes.
  An algometer Wagner FPI 10-WA will be used to determine the PPT in infraespinatus muscle.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Pecos-Martin, PhD, Study Chair — Alcala University
Locations (1):
- Clinical University Physiotherapy and pain, Alcalá de Henares, Madrid, Spain